CLINICAL TRIAL: NCT01453270
Title: Emergency Department Management of Sepsis Patients: A Goal-Oriented Non-Invasive Sepsis Trial
Acronym: AGONIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGONIST
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Sepsis; Shock, Septic
Keywords: Sepsis; Emergency medicine; Cardiac output; Stroke volume; Lactate
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NICOM and PLR (Experimental): A systematic approach to resuscitation started in the ED and using a step-wise approach to optimize cardiac preload, afterload, and contractility, thus optimizing oxygen delivery to the tissues will be applied to the intervention group using the Non-Invasive Cardiac Output Monitor (NICOM) and passive leg-raising (PLR) maneuver.
  Interventions: Device: NICOM
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Device: NICOM — Assessment of fluid responsiveness will be done using the non-invasive cardiac output monitor (NICOM) and passive leg-raising (PLR) maneuver to target mean arterial pressure of between 65mmHg and 90mmHg; and change in stroke volume index (SVI) less than 10%, prior to administration of fluid boluses.
  Arms: NICOM and PLR
Other: Usual care — Usual care is given at the clinician's discretion in accordance with current best practice. Standard treatment may involve treatment with intravenous fluids, and medications to support the blood pressure and heart.
  Arms: Usual care

SUMMARY:
The purpose of this study is to determine whether the use of a 3-hour protocol utilizing non-invasive hemodynamic optimization treatment strategy results in better outcome and lower hospital costs in patients who present with severe bloodstream infections to the Emergency Department (ED).

DETAILED DESCRIPTION:
Severe sepsis is a syndrome where the body develops organ dysfunction secondary to uncontrolled inflammatory response to infection. Various resuscitation bundles have been formulated and practised to treat severe sepsis, such as early goal-directed therapy (EGDT). EGDT involves the insertion of invasive catheters in patients with severe sepsis or septic shock using serial measurements to guide therapy and achieve hemodynamic goals, such as mean arterial pressure (MAP), central venous pressure (CVP) and central venous oxygen saturation (ScvO2) by 6 hours. The drawbacks include the invasive nature of inserting these catheters with its complications and tedium to set up the equipment. A non-invasive approach using the Non-Invasive Cardiac Output Monitor (NICOM) and passive leg raising (PLR) maneuver to guide fluid and vasoactive agent therapy targeting fluid responsiveness and MAP may be able to achieve better outcome, measured by lactate clearance at 3 hours and at a lower hospitalization cost.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of at least 2 systemic inflammatory response syndrome (SIRS) criteria
* Suspected infection
* Serum lactate ≥3mmol/L

Exclusion Criteria:

* Age below 21 years
* Known pregnancy
* Prisoners
* Do-not-attempt resuscitation status
* Known severe aortic insufficiency or severe anatomic abnormalities of the thoracic aorta
* Primary diagnosis of trauma, burns, active seizures, acute cerebral vascular accident, acute coronary syndrome, status asthmaticus, major cardiac arrhythmias, active gastrointestinal haemorrhage, seizure or drug overdose
* Requirement for immediate surgery
* Inability to do PLR (e.g. ankylosis of hip joint, severe sciatica)
* Treating physician deems aggressive care unsuitable
* Those unable to give informed consent and unable to comply with study requirements

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Lactate clearance >20% | 3 hours
  Arterial lactate levels will be measured at 0 and 3 hours to determine degree of lactate clearance at 3 hours.

SECONDARY OUTCOMES:
Total hospital cost | At discharge, death or 28 days, whichever occurs earlier

CONTACTS AND LOCATIONS:
Overall Officials: Win Sen Kuan, MBBS, Principal Investigator — National University Health System, Singapore; Irwani Ibrahim, MBBS, Principal Investigator — National University Health System, Singapore; Benjamin SH Leong, MBBS, Principal Investigator — National University Health System, Singapore; Malcolm Mahadevan, MBBS, Study Chair — National University Health System, Singapore; Yin Bun Cheung, PhD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore